CLINICAL TRIAL: NCT04660383
Title: Effects of Intradialytic Inspiratory Muscle Training at Different Intensities on Diaphragm Hypertrophy and Functional Capacity in Patients Undergoing Hemodialysis: a Randomized Clinical Trial.
Brief Title: Intradialytic Inspiratory Muscle Training at Different Intensities and Functional Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2020-0458
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Kidney Failure, Chronic
Keywords: intradialytic training; Inspiratory Muscle Training; Diaphragm Hypertrophy; Functional capacity; End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IMT 50 (Experimental): IMT intervention: IMT50 - 50% of the maximum inspiratory pressure (MIP), using equipment "Threshold IMT®" or "Power Breathe®", which are respiratory incentives of linear pressure load, where the patient uses a nose clip and breathes through a mouthpiece with a resistance in the inspiratory branch, using the respective MIPs.
  Interventions: Device: Inspiratory Muscle Training
- IMT 30 (Experimental): IMT intervention: IMT30 - 30% of the maximum inspiratory pressure, using equipment "Threshold IMT®" or "Power Breathe®", which are respiratory incentives of linear pressure load, where the patient uses a nose clip and breathes through a mouthpiece with a resistance in the inspiratory branch, using the respective MIPs.
  Interventions: Device: Inspiratory Muscle Training
- IMT 10 (Sham Comparator): IMT intervention: IMT10 - 10% of the maximum inspiratory pressure, using equipment "Threshold IMT®" or "Power Breathe®", which are respiratory incentives of linear pressure load, where the patient uses a nose clip and breathes through a mouthpiece with a resistance in the inspiratory branch, using the respective MIPs.
  Interventions: Device: Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Training — Patients will be submitted to three weekly IMT sessions in three different intensities for a period of twelve weeks, totaling 36 sessions.

SUMMARY:
Investigate the effects of Inspiratory Muscle Training (IMT) performed during hemodialysis (HD) procedures in patients with end stage kidney disease (ESKD). With intervention of thirty-six IMT sessions, performed three times a week, at an intensity of 50%, 30% and 10% (sham) of the maximum inspiratory pressure (MIP).

DETAILED DESCRIPTION:
Introduction: Chronic kidney disease (CKD), especially in its final stage (ESKD), is associated with an increased risk of cardiovascular complications and mortality. Part of this risk can be attributed to the fact that patients with ESKD adopt sedentary behavior.

Objectives: To investigate the effects of Inspiratory Muscle Training (IMT) performed during hemodialysis (HD) procedures in patients with ESKD.

Methodology: Randomized double-blind clinical trial, controlled by sham. Location: Nephrology Sector, Hospital de Clínicas de Porto Alegre (HCPA) Participants: three groups of 12 patients with ESKD on HD randomized to three IMT intensities.

Intervention: Thirty-six IMT sessions, performed three times a week, at an intensity of 50%, 30% and 10% (sham) of the maximum inspiratory pressure (Pimax).

Main outcomes: Functional capacity, diaphragm hypertrophy, respiratory muscle strength, lung volume, blood pressure and quality of life.

Statistical Analysis: Presentation of data in absolute and relative numbers, and through means and standard deviations. To compare the groups, ANOVA will be used, with significance less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients who have been on HD for at least three months;
* In physical conditions to perform the tests proposed by the study;
* With stable CKD for at least 30 days (with no hospitalization);

Exclusion Criteria:

* Patients with a recent history of arrhythmias;
* Recent hospitalization (<3 months);
* Recent acute myocardial infarction (<6 weeks);
* HD routine less than 2X / week;
* Muscle or respiratory changes (eg, chronic obstructive pulmonary disease (COPD));
* Unstable angina;
* Severe valve disease;
* Uncontrolled hypertension;
* Hemoglobin concentration <10 g / dL;
* Participation in a study with intradialytic exercise in the six months preceding this study;
* Refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Capacity (6MWT) | Baseline, 3 months
  The 6MWT is a useful, validated, and well-tolerated tool that requires no specialized equipment, used to determine the functional capacity of individuals with chronic kidney disease. 19 In addition, the 6MWT is able to represent the submaximal level of functional capacity (e.g., daily physical activity). The results will be defined as the difference in meters in distance covered at weeks 0 and 12. Participants will be instructed to walk on a flat, straight corridor, and will be told that the objective of the test is to walk as far as possible for six minutes at a self-selected speed.
Change in Functional Capacity (CPET) | Baseline, 3 months
  Patients will be submitted to CPET on an exercise bike, using an incremental loading protocol according to the guidelines published by the American Thoracic Society / American College of Chest Physicians.
Change in diaphragm hypertrophy | Baseline, 3 months
  Mode B ultrasound (EnVisor C, Philips, Bothell, Washington) with a 12.0 MHz ultrasound probe (L12-3, Philips) will be used for the image of the diaphragm in the apposition zone, the vertical section that rests against the lateral portion of the right rib cage, with the method described by Wait et al.

SECONDARY OUTCOMES:
Change in ambulatory blood pressure measurement (ABPM) | Baseline, 3 months
  ABPM is a method that allows indirect and intermittent blood pressure recordings for a period of 24 hours, while patients perform their daily life activities.
Change in respiratory muscle strength | Baseline, 3 months
  Maximal Inspiratory Measure and Maximal Expiratory Measure: will be carried out by GlobalMed® MVD300 manovacuometry equipment.
Quality of Life assessed by KDQoL Short-Form | Baseline, 3 months
  Assessed by Kidney Disease Quality of Life Short-Form

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira MS, Ferrari F, Dipp T, Carvalho G, Bitencourt EDS, Saffi M, Stein R. Effects of intradialytic inspiratory muscle training at different intensities on diaphragm thickness and functional capacity: clinical trial protocol in patients undergoing haemodialysis. BMJ Open. 2023 Jan 27;13(1):e066778. doi: 10.1136/bmjopen-2022-066778. PMID 36707111